CLINICAL TRIAL: NCT04493359
Title: Switch or Maintenance of Renin-Angiotensin System Inhibitors in Patients With Covid-19: A Randomized Proof of Concept Trial
Brief Title: Switch of Renin-Angiotensin System Inhibitors in Patients With Covid-19
Acronym: SWITCH-COVID
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Dificulteis in enrolling patients
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Caramelli, MD. PHD., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33575220.9.0000.0068
Record Dates: First submitted 2020-07-29; First posted 2020-07-30 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Angiotensin II Receptor Antagonist Adverse Reaction
Keywords: covid19; ace inhibitors; ace2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Switch therapy (Experimental): Renin-angiotensin system inhibitors will be changed for other anti-hypertensive classes.
  Interventions: Drug: Renin-angiotensin system inhibitors
- Maintenance therapy (No Intervention): Renin-angiotensin system inhibitors will be kept during in-hospital stay

INTERVENTIONS:
Drug: Renin-angiotensin system inhibitors — switch anti-hypertensive class
  Arms: Switch therapy

SUMMARY:
The SWITCH-COVID trial will randomize patients with COVID-19 that are currently using renin-angiotensin system inhibitors for treating hypertension to maintain the therapy during in-hospital stay or switch the therapy to other antihypertensive classes.

DETAILED DESCRIPTION:
Patients eligible for the study, after signing informed consent will be randomized 1:1 for maintenance of renin-angiotensin system inhibitors or switching the antihypertensive therapy for other classes according to a pre-specified protocol.

Patients are going to be followed during hospital stay for evaluation of clinical endpoints. Also blood and urine samples will be acquired for evaluation of renin-angiotensin system activation.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension in use of renin-angiotensin system inhibitors
* Confirmed COVID-19 infection by rt-PCR, serology tests or typical clinical presentation and chest CT.
* Symptoms onset < 96h
* Need for hospitalization

Exclusion Criteria:

* Heart failure
* Previous cerebrovascular disease
* Previous myocardial infarction
* Blood pressure > 180 x 100 mmHg
* Need for 3 or more anti-hypertensive classes
* Use os spironolactone
* Severe pulmonary disease
* Contraindication for using other anti-hypertensive classes (calcium channel blockers, hydralazine, diuretics or nitrates)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Need for ICU or mortality | 30 days
  Combined of need for ICU or mortality

SECONDARY OUTCOMES:
High sensitivity troponin levels and covid-19 severity | 30 days
  Evaluate correlation between hs-TnT and covid-19 severity
ACE-2 activity and disease severity | 30 days
  Evaluate correlation of ACE-2 activity and disease severity
ACE-2 activity with different Renin-angiotensin system inhibitors | 30 days
  Evaluate correlation of ACE-2 activity and Renin-angiotensin system inhibitors
Blood control and acute renal failure | 30 days
  Evaluate blood pressure control and acute renal failure in each arm (safety)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - Incor HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Data may be requested for collaboration projects